CLINICAL TRIAL: NCT05942521
Title: Effects of Subconscious Memory Extinction in Patients With Alcohol Dependence and Its Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Kangning Hospital (Other)
Responsible Party: Principal Investigator, Xiaojian Jia, Professor, Shenzhen Kangning Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-K013-01
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol; Craving; Extinction training; Subconscious
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Very brief extinction (Experimental): Enrolled participants would receive very brief extinction approximately 25 minutes per day for 2 days.
  Interventions: Behavioral: Very brief extinction
- Very brief neutral extinction (Sham Comparator): Enrolled participants would receive very brief neutral extinction for approximately 25 minutes per day for 2 days.
  Interventions: Behavioral: Very brief neutral extinction
- Clearly visible extinction (Active Comparator): Enrolled participants would receive clearly visible extinction therapy for approximately 25 minutes per day for 2 days.
  Interventions: Behavioral: Clearly visible extinction

INTERVENTIONS:
Behavioral: Very brief extinction — The very brief extinction presents a very short (33ms) repetitive sequence of alcohol cues, followed by a "masking" stimulus(117ms), which masks the alcohol cues. In the case of repeated exposure to alcohol stimulation, the response to the stimulation is desensitized at the level of unconscious processing.
  Arms: Very brief extinction
Behavioral: Clearly visible extinction — The clearly visible extinction presents a repetitive sequence of alcohol cues(150ms) without a "masking" stimulus. In the case of repeat exposure to alcohol stimulation, the response to the stimulation is desensitized at the level of conscious processing.
  Arms: Clearly visible extinction
Behavioral: Very brief neutral extinction — The very brief neutral extinction presents a very short (33ms) repetitive sequence of neutral cues, followed by a "masking" stimulus(117ms), which masks the neutral cues. In the case of repeated exposure to neutral stimulation, the response to the stimulation is desensitized at the level of unconscious processing.
  Arms: Very brief neutral extinction

SUMMARY:
In this study, the subconscious memory extinction therapy based on very brief exposure is used to intervene to reduce the alcohol craving of alcohol-dependent patients, prevent relapse, and observe the psychological craving, heart rate, skin conductance, and pupil diameter changes of the patients during the brief exposure extinction. The main questions it aims to answer are:

1. Whether subconscious extinction intervention would reduce psychological craving and alcohol relapse?
2. What is the mechanism of subconscious extinction intervention in alcohol dependence?

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period to determine eligibility for study entry. patients who meet the eligibility requirements will be randomized in very brief extinction, clearly visible extinction, or very brief neutral extinction. This study will recruit alcohol-dependent participants aged 18-60 in the ward, observe reported subjective scores during the extinction, and record the heart rate, skin conductance, pupil diameter, and ERP changes.

ELIGIBILITY:
Inclusion Criteria:

1. Adopt DSM-IV alcohol dependence diagnostic criteria;
2. Complete detoxification treatment without obvious withdrawal symptoms;
3. Informed consent, voluntary participation.

Exclusion criteria:

1. Acute alcohol dependence withdrawal period;
2. Patients who meet the DSM-Ⅳ diagnosis of psychoactive substances or non-psychoactive substances other than alcohol (except nicotine);
3. Previous acceptance experienced similar exposure therapy;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in alcohol craving by using Visual Analog Scale of Alcohol Craving at week 1. | baseline and week 1
  Alcohol-specific Visual Analog Scale is a valid measurements of craving for a alcohol. Possible scores range from 0(no craving) to 10 (want to drink imediately). Change= (week 1 score - baseline score)
Relapse rate | Four week after intervention
  Percentage of participants who relapse by assuming that drinking alcohol on more than 3 days in a month in anunrestricted environment is re-drinking

SECONDARY OUTCOMES:
Skin conductance level (SCL) | During the intervention period
  Thus skin conductance level can serve as a stable and useful index of autonomic arousal in clinical trials. Skin conductance signals are measured via electrodes placed on fingertips, arrange from 0 to 50 uS.
Pupil diameter | During the intervention period
  The pupil diameter is measured by Eyelink 1000 plus eyetracking, Pupil size data are available with every data point collected by the EyeLink 1000 Plus. To evaluate the level of accuracy obtained in pupil size measures, dots between 2.0 and 5.0 mm in diameter were laser printed.
Event-relatred potential (ERP) | During the intervention period
  An ERP is a technique that can be used to assess how the brain is functioning in response to stimulation. Event-related potentials (ERPs) are derived from electroencephalographic (EEG) measurement of neural activity. The 64-channel EEG system from Brain Products company would be used to measure P300, N400, and slow potential.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojian Jia, Principal Investigator — Shenzhen Kangning Hospita
Locations (1):
- Shenzhen Kangning Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No